CLINICAL TRIAL: NCT04881526
Title: Ketone Ester Supplementation on Neuro-cardiovascular Responses to Stress in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Philip Millar, Associate Professor, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 21-02-019
Record Dates: First submitted 2021-05-05; First posted 2021-05-11 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Ketosis
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone ester drink (Active Comparator)
  Interventions: Dietary Supplement: D-beta-hydroxybutyrate
- Placebo drink (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: D-beta-hydroxybutyrate — Drink containing D-beta-hydroxybutyrate administered at a dose of 395 mg/kg.
  Arms: Ketone ester drink
Dietary Supplement: Placebo — Isocaloric flavored water with medium-chain triglyceride oil.
  Arms: Placebo drink

SUMMARY:
Ketone ester supplementation has become increasingly popular as an athletic supplement. However, the metabolic effects of these supplements on exercise performance are controversial. One potential reason for lack of an ergogenic benefit could be the effects of ketone bodies on other bodily systems, such as the sympathetic nervous system. During exercise and stress the body increases the activity of the sympathetic nervous system. This causes blood vessels to constrict (get smaller) and can increase blood pressure. Studies have shown that ketone bodies can suppress the sympathetic nervous system in mice. Additionally, ketone ester supplementation can reduce blood pressure in healthy adults. In humans, direct measures of sympathetic activity are usually made from sympathetic outflow to muscle, also called muscle sympathetic nerve activity (MSNA). Using a ketone ester supplement, the investigators plan to measure blood pressure and sympathetic outflow to muscle at rest and during handgrip exercise and a mathematical task stress test to investigate the effect of ketones on neuro-cardiovascular stress responses.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 40 years of age
* Healthy, free of known cardiovascular, metabolic, or musculoskeletal disease

Exclusion Criteria:

* History of smoking (within 3 months), diagnosed cardiovascular or metabolic disease, recent musculoskeletal injury preventing handgrip exercise, prescription of chronic medications other than oral contraceptives.
* Current or recent (within 6 months) use of ketone ester supplementation or participation in a ketogenic diet.
* Inability to abstain from drugs, caffeine, alcohol, or strenuous physical activity prior to the study visit.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Muscle sympathetic nerve activity | Baseline - Immediately before active and control interventions
  Microneurography of fibular nerve
Muscle sympathetic nerve activity | Post-intervention - Immediately following active and control interventions
  Microneurography of fibular nerve
Blood pressure | Baseline - Immediately before active and control interventions
  Finger plethysmography
Blood pressure | Post-intervention - Immediately following active and control interventions
  Finger plethysmography

SECONDARY OUTCOMES:
Forearm blood flow | Baseline - Immediately before active and control interventions
  Brachial artery Doppler ultrasound
Forearm blood flow | Post-intervention - Immediately following active and control interventions
  Brachial artery Doppler ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Philip Millar, PhD, Principal Investigator — University of Guelph
Locations (1):
- University of Guelph - Human Cardiovascular Physiology Laboratory, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No